CLINICAL TRIAL: NCT00773435
Title: Assessing the in Vivo Effect of Echinacea Purpurea on Markers of Immune Activities in Children
Brief Title: Effects of Echinacea in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided to conduct study in adults first
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, James Taylor, Professor, Pediatrics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: A41256; 5U01AT002400 (NIH)
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2008-12

CONDITIONS: Upper Respiratory Infections
Keywords: Upper respiratory tract infections; Children; Echinacea; Prevention; Immune modulation
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Echinacea extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Echinacea purpurea (Active Comparator)
  Interventions: Biological: Echinacea purpurea 100 mg/ml in liquid formulation
- 2. placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: Echinacea purpurea 100 mg/ml in liquid formulation — 10 ml BID for 10 consecutive days at the start of 3 consecutive 30 day periods
  Arms: 1. Echinacea purpurea
Other: placebo — 10 ml PO BID for 10 consecutive days at the beginning of 3 consecutive 30 day periods
  Arms: 2. placebo

SUMMARY:
The goal of the this study is to determine if Echinacea purpurea stimulates the immune system in children. For the study, 40 healthy children, 6-11 years old will be randomized to receive Echinacea purpurea or placebo for 10 days in 3 consecutive months. Blood samples will be obtained in the children just before starting study medication, during the first course of medication and either just prior to starting the second course of medication or 50 days following the last of the three courses of medication. Markers of immune activity in children receiving Echinacea or placebo will be compared.

DETAILED DESCRIPTION:
This is an application to study the biologic activity of a specific formulation of Echinacea purpurea in children 6-11 years old. The goal of the study is to determine if Echinacea purpurea is associated with activation of immune markers including cytokines such as tumor necrosis factor alpha (TNF), interferon alpha, interferon gamma, and interleukins 2, 6, and 12 (IL-2, IL-6, and IL-12), as well CD25 and CD69 activation. A total of 40 study children will be randomized to receive either the Echinacea purpurea formulation or placebo for 10 consecutive days at the start of 3 consecutive 30-day periods. Blood samples will be obtained at baseline, at the time of "peak" TNF activity, and either 30 or 120 days after beginning the study medication. Prior to beginning this pediatric study "peak" TNF activity will be determined by administering the Echinacea purpurea to 3 adult volunteers for 10 days and doing frequent blood sampling during this period. If it is demonstrated that this formulation of E purpurea has biologic activity, a large randomized controlled trial is planned to determine if E purpurea can prevent upper respiratory tract infection (URI) in children 2-11 years old.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 6-11 years old
* Parent/Caregiver who can read and speak English
* One child per family

Exclusion Criteria:

* History of allergic reaction to Echinacea or related species
* History of asthma
* History of allergic rhinitis
* History of autoimmune disease

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
TNF levels | During first course of study medication

SECONDARY OUTCOMES:
CD25/CD69 activation | 120 days
IL-2, IL-6, IL-12, interferon alpha, interferon gamma, TNF levels | 120 days
specific and general adverse events | 120 days

CONTACTS AND LOCATIONS:
Overall Officials: James A Taylor, Principal Investigator — University of Washington